CLINICAL TRIAL: NCT03549546
Title: Expression of the Inhibitory Receptors on Lymphocytes T Cells After Lung Cancer Surgery.
Acronym: POIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1708182; 2017-A03391-52 (Other: ID-RCB)
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2018-12

CONDITIONS: Lung Cancer; Surgery
Keywords: Lymphopenia; Lung cancer surgery; TIM-3; PD-1; CTLA-4; lymphocytes; CD4; CD8
MeSH Terms: conditions — Lung Neoplasms; Lymphopenia; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing lung cancer surgery (Other): Patients undergoing lung cancer surgery will be included. Blood samples will be collected.
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — Blood samples will be collected in patients undergoing lung cancer surgery:
  * before lung cancer surgery,
  * the next day lung cancer surgery,
  * 3 days after lung cancer surgery. They will be treated in flow cytometry.

SUMMARY:
Postoperative pneumonia is one of the most common complications after lung cancer surgery and associated with a morbidity and mortality. Postoperative lymphopenia has been recently identified as one of risk factors for postoperative pneumonia. According to recent studies in polytrauma, cancer or septic shock, T cells dysfunction may be related to high expression of inhibitory receptors on lymphocytes.

DETAILED DESCRIPTION:
This study will investigate prospectively TIM-3, PD-1 and CTLA4 expression on lymphocytes T cells before and after lung cancer surgery. Patients ≥ 18 years with no history of immunosuppressive state will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years undergoing lung cancer surgery by thoracoscopy

Exclusion Criteria:

* Patient under guardianship/curatorship
* Patient who received of radiotherapy or chemotherapy in the last 6 months
* Patient under immunosuppressive treatment or dose of corticoids over 10 mg/day prednisolone or equivalent
* Patient with history of malignant blood disease or auto-immune disease
* Patient suffering from HIV infection and
* Patients with pre-operative infection
* Patient with an empiric antibiotic therapy introduced at operating room

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
PD-1, TIM-3, CTLA4 on CD4/CD8 lymphocytes | Days 0, 1, 3
  Correlation between expression of PD-1, TIM-3, CTLA4 on CD4/CD8 lymphocytes and the occurrence of lymphopenia.
  Measured by blood sample before lung cancer surgery, the next day lung cancer surgery and 3 days after lung cancer surgery. Analyzed by multicolour immunolabelling in flow cytometry

SECONDARY OUTCOMES:
functionality of CD4/CD8 lymphocytes and production of IF gamma, TNF and IL-2 | Days 0, 1, 3
  Correlation between functionality of CD4/CD8 lymphocytes and production of interferon (IF) gamma, Tumor Necrosis Factor (TNF) and interleukine (IL-2).
  Measured by blood sample before lung cancer surgery, the next day lung cancer surgery and 3 days after lung cancer surgery. Analyzed by multicolour immunolabelling in flow cytometry
pneumonia | Days 3
  To analyse the occurrence of postoperative pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Dupont, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No